CLINICAL TRIAL: NCT06176885
Title: Efficacy and Safety of Camrelizumab Combined With Irinotecan, Leucovorin and Fluorouracil (FOLFIRI) Chemotherapy and Bevacizumab Targeted Induction Therapy in the First-line Treatment of Microsatellite Stable (MSS) Initially Unresectable Metastatic Colorectal Cancer: a Prospective, Multicenter, Single-arm Study
Brief Title: Efficacy and Safety of Combined With Immunotherapy After Induction Therapy With Chemotherapy and Targeted Therapy in the First-line Treatment of Microsatellite Stable (MSS) Initially Unresectable Metastatic Colorectal Cancer
Acronym: FOBECAMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: yue junhan (Other)
Responsible Party: Sponsor-Investigator, yue junhan, Director, Jinhua Central Hospital
Organization: Jinhua Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 321000
Record Dates: First submitted 2023-12-09; First posted 2023-12-20 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Hepatopulmonary metastasis; Camrelizumab; MSS; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab Group (Experimental): Combined with Camrelizumab after irinotecan leucovorin and fluorouracil (FOLFIRI) chemotherapy and bevacizumab targeted induction therapy
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Combination therapy with Camrelizumab monoclonal antibody will be administered after the initial two cycles of induction therapy.

SUMMARY:
The goal of this clinical trial is to explore the feasibility of a new mode of chemotherapy and bevacizumab induction therapy combined with immunotherapy as first-line treatment for patients with initially unresectable metastatic colorectal cancer (MSS). The main questions it aims to answer are:

1. To explore the efficacy and safety of this treatment mode
2. Try to study treatment benefit the characteristics of the crowd Participants will combined with immunotherapy after chemotherapy and bevacizumab induction therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study signed the informed consent and had good compliance
2. Body weight ≥40kg
3. Metastatic colorectal cancer confirmed by histology and/or cytology and initially unresectable
4. Microsatellite instable (MSS) or proficient Mismatch Repair (pMMR)
5. Patients have at least one measurable lesion (RECIST 1.1)
6. Eastern Cooperative Oncology Group Physical Status (ECOG PS) 0-1
7. Expected survival ≥12 weeks
8. Blood testing (not corrected with granulocyte colony-stimulating factor or other hematopoietic stimulating factor within 7 days prior to laboratory testing if not transfused within 14 days)
9. Women of reproductive age had to have a serum pregnancy test with a negative result within 14 days before treatment and be willing to use a medically approved effective contraceptive during the study and for 3 months after the last dose of study medication
10. Age 18-75 years old (including 18 and 75 years old)

Exclusion Criteria:

1. The patient had received radiation therapy surgery chemotherapy immune or molecular-targeted therapy or other investigational drugs within 4 weeks before treatment
2. An active autoimmune disease requiring systemic therapy (i.e., disease-modifying medications, corticosteroids, or immunosuppressive agents) had occurred within the previous 2 years. Replacement therapies, such as thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency, are not considered systemic treatments
3. Immunodeficiency was diagnosed within 7 days before the first treatment or received systemic steroid therapy or any other form of immunosuppressive therapy. Physiological doses of corticosteroids could be approved after consultation with the sponsor
4. She had previously received anti-vascular small molecule targeted drug therapy, such as Fruquintinib
5. Prior treatment with an irinotecan-based chemotherapy regimen
6. Symptomatic brain or meningeal metastases
7. Left colon cancer with wild-type rat sarcoma virus gene (RAS)
8. MSI-H or dificient Mismatch Repair (dMMR) metastatic colorectal cancer
9. Serious infection (e.g., intravenous antibiotic, antifungal, or antiviral) within 4 weeks before treatment, or unexplained fever > 38.5 ° C during screening/first dose
10. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
11. The patient had obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, melena, hematochezia), hemoptysis (fresh blood > 5 mL within 4 weeks), etc. Or treatment for a venous/venous thrombotic event within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism Long-term anticoagulation with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) may be required
12. At the time of screening, tumors were found to invade large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava, which were judged by the investigator to have a high risk of bleeding
13. "Active heart disease, including myocardial infarction, severe/unstable angina, occurred 6 months before treatment." Echocardiography showed that the left ventricular ejection fraction was less than 50% and the arrhythmia was not well controlled
14. Patients with other malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within the past 5 years or at the same time
15. Known allergy to the study drug or any of its excipients
16. Severe, active or uncontrolled infection
17. Any other medical condition, clinically significant metabolic abnormality, physical examination abnormality, or laboratory abnormality, a disease or condition for which there is reason to suspect that the patient is not suitable for use of the study drug (e.g., having seizures requiring treatment), or a condition that would affect interpretation of the study results, or that would place the patient at high risk, in the investigator's judgment
18. If urine routine test showed urinary protein ≥2+ and 24-hour urinary protein quantitation >1.0g

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
PFS（Disease-free Survival） | 11.5 months
  Disease-free Survival

SECONDARY OUTCOMES:
ORR（Objective Remission Rate） | 2 years
  Objective Remission Rate
Conversion resection rate | 2 years
  Conversion resection rate
OS（Overall Survival） | more than 2 years
  Overall Survival
Incidence of Treatment-Emergent Adverse Events | 2 years
  Treatment-Emergent Adverse Events，such as bleeding，thrombocytopenia，abnormal liver function，proteinuria，hypertension and so on
DCR（Disease control rate） | 2 years
  Disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery, Affiliated Jinhua Hosptial, Zhejiang University, Jinhua, Zhejiang, China